CLINICAL TRIAL: NCT03624010
Title: Open-Label Rollover Study of Levosimendan in Patients With Pulmonary Hypertension With Heart Failure and Preserved Left Ventricular Ejection Fraction (PH-HFpEF)
Brief Title: Open-Label Rollover Study of Levosimendan in PH-HFpEF Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tenax Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TNX-LVO-05
Record Dates: First submitted 2018-07-24; First posted 2018-08-09 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Hypertension Pulmonary Secondary Heart Failure; Right Sided Heart Failure With Normal Ejection Fraction; Heart Failure With Normal Ejection Fraction
MeSH Terms: interventions — Simendan

STUDY DESIGN:
Intervention Model Description: Open-label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Levosimendan (Experimental): A sterile 2.5 mg/mL concentrate solution that is diluted in 5% Dextrose or 0.9 Normal Saline to achieve a 50 microgram/min solution for infusion
  Interventions: Drug: Levosimendan 2.5 mg/ml Injectable Solution

INTERVENTIONS:
Drug: Levosimendan 2.5 mg/ml Injectable Solution — A sterile 2.5 mg/mL concentrate solution that is diluted in 5% Dextrose or 0.9 Normal Saline to achieve a 50 microgram/min solution for infusion

SUMMARY:
PH-HFpEF patients will receive weekly open-label doses of levosimendan and be periodically evaluated for safety and effectiveness in extended use.

DETAILED DESCRIPTION:
This study will enroll PH-HFpEF patients that have completed a controlled levosimendan study. These patients will receive weekly open-label doses of levosimendan and be periodically evaluated for safety and effectiveness in extended use.

ELIGIBILITY:
Inclusion Criteria:

1. Provide a personally signed and dated informed consent document prior to initiation of any study-related procedures that are not considered standard of care.
2. Completed double-blind therapy in a PH-HFpEF clinical study sponsored by Tenax Therapeutics, Inc.
3. May, in the opinion of the Investigator, benefit from continued levosimendan treatment.
4. Female patients of childbearing potential must agree to use a highly effective method of contraception.
5. Willingness and ability to comply with scheduled visits, treatment plan, laboratory tests and other study procedures.

Exclusion Criteria:

1. Discontinued treatment in the parent study for any reason other than study completion or Sponsor termination of the study.
2. Pregnant or breastfeeding women.
3. Local access to commercially available levosimendan
4. Inability to comply with planned study procedures
5. Patients with scheduled lung or heart transplant or cardiac surgery
6. Dialysis developed since enrollment in parent study (either hemodialysis, peritoneal dialysis, continuous venovenous hemofiltration, or ultrafiltration)
7. Estimated glomerular filtration rate (eGFR) <30 mL/min/1.73m2
8. Liver dysfunction with Child Pugh Class B or C (see Attachment 2)
9. Evidence of systemic bacterial, systemic fungal, or viral infection refractory to treatment
10. Weight >150kg
11. Systolic blood pressure (SBP) cannot be managed to ensure SBP >100 mmHg at initiation of study drug
12. Heart rate >100 bpm with study drug, persistent for at least 10 minutes at screening.
13. Hemoglobin < 80 g/L
14. Serum potassium < 3.0 mmol/L or > 5.5 mmol/L at baseline that is unresponsive to management

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-11-14 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-02-01 (Actual)

PRIMARY OUTCOMES:
Clinical Safety measured by number of adverse events (AEs ) | 2 years
  Long-term safety profile of levosimendan measured by number of adverse events (AEs )

SECONDARY OUTCOMES:
6-minute walk test (6MWT) | 2 years
  Exercise capacity, measured as a distance traveled in 6 minutes
Patient global assessment | 2 years
  Patient's assessment of well-being, based on a six-point Likert scale (1 =worst, 5= best)
Physician's Assessment of Functional Class | 2 years
  Physician's Assessment of New York Heart Association (NYHA) Classification (one of four categories based on how much the patient is limited during physical activity. (Class I, no limitation of physical activity to Class IV, marked limitation of physical activity)
Clinical Events: Death and hospitalizations | 2 years
  Incidence of death or hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Stuart Rich, MD, Principal Investigator — Tenax Therapeutics, Inc.
Locations (9):
- United States (9):
  - Stanford Healthcare, Stanford, California
  - Northwestern Memorial Hospital, Chicago, Illinois
  - University of Minnesota Medical Center, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - UPMC Presbyterian Hospital, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - UW Health University Hospital, Madison, Wisconsin